CLINICAL TRIAL: NCT02662491
Title: Effects of Vitamin D and Calcium Supplementation on Health of UAE Citizens
Brief Title: Effects of Vitamin D and Calcium Supplementation on Health and Well-being of Vitamin D Deficient UAE Citizens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Salah Gariballa, Professor, United Arab Emirates University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/05; VITD (Other: UAEU)
Record Dates: First submitted 2016-01-13; First posted 2016-01-25 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Calcium

STUDY DESIGN:
Intervention Model Description: Calcium 600mg, vitamin D 2000IU, both or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- vitamin D and calcium (Experimental): daily oral vitamin D(3) (2000 IU) and calcium (600 mg) for 6 months
  Interventions: Dietary Supplement: Vitamin D and calcium
- Calcium supplement (Experimental): daily oral calcium (600 mg) for 6 months
  Interventions: Dietary Supplement: Calcium
- vitamin D supplement (Experimental): daily oral vitamin D(3) (2000 IU) for 6 months
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): daily placebo tablet for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D and calcium
  Arms: vitamin D and calcium
Dietary Supplement: Vitamin D
  Arms: vitamin D supplement
Dietary Supplement: Calcium
  Arms: Calcium supplement
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The trial plan to determine whether a daily capsule containing vitamin D(3) (2000 IU), calcium (600 mg), both, or a placebo for 6 months in UAE citizens with evidence of vitamin D deficiency will lead to a clinical benefit. The proposed study will also determine the threshold of vitamin D and calcium intake or levels considered optimal for UAE citizen's health

DETAILED DESCRIPTION:
The proposed study is a two by two factorial, randomized controlled intervention trial. Following informed written consent of eligible subject's blood and urine samples will be taken for measurements of vitamin D, markers of bone turnover and related biochemical variables. Patients who have evidence of vitamin D deficiency will then be randomly assigned to receive daily vitamin D(3) (2000 IU), calcium (1000 mg), both, or a placebo for 6 months. All subjects will have a calcium and vitamin D rich food and other lifestyle modification advises during the study period. Patients will otherwise be managed according to standard practice. Clinical assessment that includes general and self-rated health, bone density, muscle strength, physical activity and dietary intakes will be performed at baseline, and repeated at 3, 6 and 12 months post-randomisation.

Information on other important variables likely to influence vitamin D status including age, reproductive & menopausal history, smoking, medications, adiposity, exposure to sunlight, dietary intake including supplements, skin pigmentation, chronic illness and medications will be collected and adjusted for during the analysis

ELIGIBILITY:
Inclusion Criteria:

1. biochemical evidence of vitamin D deficiency

Exclusion Criteria:

1. renal disease or stones or hypercalcaemia,
2. Use of calcium and/or vitamin D supplementation, bisphosphonates, steroid medications, hormones or diuretics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Muscle pains | 6 months
  Muscle pains measured using a questionnaire
Muscle strength | 6 months
  Muscle strength measured using dynamometer
Vitamin D level | 6 months
  vitamin D level measured using liquid chromatography

SECONDARY OUTCOMES:
Dietary vitamin D intake | 6 months
  dietary vitamin D intake assessed by a food frequency questionnaire
Dietary calcium intake | 6 months
  Dietary calcium intake assessed by a food frequency questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine & Health Science, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gariballa S, Yasin J, Alessa A. A randomized, double-blind, placebo-controlled trial of vitamin D supplementation with or without calcium in community-dwelling vitamin D deficient subjects. BMC Musculoskelet Disord. 2022 May 3;23(1):415. doi: 10.1186/s12891-022-05364-z. PMID 35505326